CLINICAL TRIAL: NCT04717960
Title: Evaluation Of Role Of Platelet Rich Plasma In Treatment Of Patients Suffering From Atrophic Rhinitis
Brief Title: Evaluation of Efficacy of Platelet Rich Plasma as Anew Modality for Treatment of Atrophic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Saad Badry Abaas, Evaluation Of Role Of Platelet Rich Plasma In Treatment Of Patients Suffering From Atrophic Rhinitis, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-21-01-07
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Atrophic Rhinitis
Keywords: Atrophic rhinitis
MeSH Terms: conditions — Rhinitis, Atrophic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group group (1) (Active Comparator): the group which will undergo submucosal injection of platelet rich plasma
  Interventions: Procedure: nasal submucosal injection of platelet rich plasma
- comparative group group (2) (No Intervention): patients using the usual lines of medical treatment like nasal douching and lubricants

INTERVENTIONS:
Procedure: nasal submucosal injection of platelet rich plasma — * The selected region will be inﬁltrated with a cold saline solution with addition of 1 mL of adrenaline and 25 mL of 2% lignocaine per 500 mL saline.
  * Platelet-rich plasma is prepared by drawing 10 mL of blood sample from the patient.
  * The blood will be centrifuged at 1530 g for 10 min to obtain platelet-poor plasma.
  * This will again centrifuged at 2720 g for 10 min to get platelet-rich plasma.
  * Approximately 1 mL of platelet-rich plasma will be obtained from 10 mL blood. Usually amount of about 3ml is needed to be injected in each nostril at the affected sites of inferior and middle turbinates, septum and floor of the nose. Platelet rich plasma injected into the affected area after degranulating the platelet by adding 0.5 mL of calcium chloride.
    * Injection interval of 2 weeks (up to total 3 consecutive injections).
    * Follow-up duration: 4 months
  Arms: study group group (1)

SUMMARY:
An interventional hospital based study will be undertaken from February 2021 to February 2023 in order to determine the efficacy of platelet rich plasma as a new modality for treatment of patients suffering from atrophic rhinitis in Sohag university hospital.

DETAILED DESCRIPTION:
* Random sample will be taken from patients presenting with atrophic rhinitis to ear, nose and throat outpatient clinic in Sohag University Hospital during the period extending from February 2021 to October 2022 (taking in consideration the follow up time of the last case which will take four months). Patients will be divided randomly into two groups. The division of patients subjected to treatment will be obtained by a random sequence of computer generated numbers. One group will be subjected to submucosal platelet-rich plasma (PRP) injection (study group) and the other group will be subjected to the usual conservative lines of treatment including nasal douchings, frequent local care and mucosal lubricants (control group).

All patients will be subjected to:

1. Full history taking and clinical examination.
2. Symptom score, sinonasal outcome test-25 (SNOT 25) will be noted at the beginning and after treatment.
3. Diagnostic nasal endoscopy and the results will be noted under four objective variables; these will be noted and the scores at the beginning and the end of 12 weeks of therapy will be statistically compared in both groups; 1. Crusting (nil = 0, minimal=1, gross = 2) 2. Status of nasal mucosa (normal = 0, congested = 1, Pale Atrophic which often indicative of underlying squamous metaplasia =2) 3. Nature of secretions (thin = 0, thick = 1) 4. Condition of nasal cavity (normal size = 0, roomy (see nasopharynx) = 1)
4. Routine Laboratory investigation: looking for iron deﬁciency anemia, thrombocytopenia.
5. Baseline nasal biopsy and only those with histopathological features of atrophic rhinitis will be included in the study. Five subheadings for histopathology; Each variable was assigned a score of 0, 1 or 2 where 0 representing normal nasal mucosal features whereas 2 signifying extreme variation, the biopsy will be repeated after 12 weeks of treatment;

<!-- -->

1. Status of epithelium: respiratory epithelium (pseudo stratified columnar ciliated epithelium, squamous metaplasia (partial/total ± keratinization); Denuded or not
2. Status of mucous (goblet) cells (Normal glands / ↓ number and size / Absence)
3. Condition of blood vessels (Reduced vascularity or Dilated blood vessels / Periarteritis/ Endarteritis).
4. Tunica propria:

   Granulation tissue Presence of Chronic inﬂammatory cellular inﬁltrate Degree of Fibrosis Chronic inﬂammatory cellular inﬁltration with ﬁbrosis Basement membrane (Normal / Ill-deﬁned /Thickened) Seromucinus glands especially the serous component. 6-Assess the nasal mucociliary function using saccharin test (primary outcome at beginning of study): The test will be done at the commence of the study and 12 weeks later on. A score of 0-1 is given to time lag where (0; normal: 1; prolonged).

   First group will be treated with nasal submucosal platelet rich plasma injection as follows; • The selected region will be inﬁltrated with a cold saline solution with addition of 1 mL of adrenaline and 25 mL of 2% lignocaine per 500 mL saline.
   * Preparation of PRP:
   * Platelet-rich plasma is prepared by drawing 10 mL of blood sample from the patient.
   * The blood will be centrifuged at 1530 g for 10 min to obtain platelet-poor plasma.
   * This will again centrifuged at 2720 g for 10 min to get platelet-rich plasma.
   * Approximately 1 mL of platelet-rich plasma will be obtained from 10 mL blood. Usually amount of about 3ml is needed to be injected in each nostril at the affected sites of inferior and middle turbinates, septum and floor of the nose. Platelet rich plasma injected into the affected area after degranulating the platelet by adding 0.5 mL of calcium chloride.
   * Injection interval and follow-up duration o Injection interval of 2 weeks (up to total 3 consecutive injections).

     o Follow-up duration: 4 months.
   * Patients will be discharged from the hospital next day with oral antibiotics and anti-inﬂammatory agents for 1 week.

   Second group acting as a control, will be treated over a period of 4 months only with alkaline nasal douching and mucosal lubricants one -three times daily.

   • Patients will be followed-up at intervals of 2-4 weeks post-therapy for a period of 4 months. Observation items, clinical assessment items and evaluation method will be statistically compared:

1. Access the nasal mucosal status using diagnostic nasal endoscopy; monthly and at the end of therapy.

2. Nasal mucocilirary flow rate by Saccharine test; once per month. 3. Fill in the nasal symptom scores using Nasal Obstruction Symptom Evaluation (NOSE) Instrument, SNOT- 25 monthly.

4. The nasal biopsy will be repeated in all cases at the end of 12-week therapy and the results will be noted under same variables and scored in the same manner. The scores at the beginning of the therapy and at 12 weeks, will be statistically compared.

*All demographic data of the patients will be collected, analyzed and presented using SPSS version 21. Appropriate statistical tests will be used for comparing the results and statistical significance for each item between both groups of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary atrophic rhinitis
* patients with empty nose syndrome

Exclusion Criteria:

* patients with secondary atrohic rhinitis except for those with empty nose syndrome
* patients with bleeding disorders mainly platelet disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Degree of change in histopathological pattern of nasal mucosa | 12 weeks after end of the procedure.
  A nasal mucosal biopsy will be obtained in all cases. Five subheadings for histopathology; Each variable was assigned a score of 0, 1 or 2 where 0 representing normal nasal mucosal features, whereas 2 signifying extreme variation,
  1. Status of epithelium: respiratory epithelium (pseudo stratified columnar ciliated epithelium, squamous metaplasia (partial/total ± keratinization); Denuded or not
  2. Status of mucous cells (Normal glands / ↓ number and size / Absence)
  3. Condition of blood vessels (Reduced vascularity or Dilated blood vessels / Periarteritis/ Endarteritis).
  4. Tunica propria:
  Granulation tissue Presence of Chronic inﬂammatory cellular inﬁltrate Degree of Fibrosis Chronic inﬂammatory cellular inﬁltration with ﬁbrosis Basement membrane (Normal / Ill-deﬁned /Thickened) Seromucinus glands especially the serous component
Degree of change in patient satisfaction and quality of life | 12 weeks after end of the procedure.
  Symptom score, Sinonasal Outcome Test 25 (SNOT 25) will be noted .

SECONDARY OUTCOMES:
Assess the nasal mucociliary function . | 12 weeks after end of the procedure.
  using saccharin test 0.5 mm sized particle will be placed approximately 1 cm behind the anterior end of inferior turbinate in sitting position with the head flexed about 10 degrees to avoid particle falling back into nasopharynx. The patient will be asked to swallow after every 50 seconds and not to sniff or drink. He/she will be asked to tell immediately when gets sweet taste of saccharine. The time elapsing until the first experience of sweet taste will be recorded as nasal mucocilliary flow rate. The test will be done at the commence of the study and 12 weeks later on. A score of 0-1 is given to time lag where (0; normal: 1; prolonged).

CONTACTS AND LOCATIONS:
Overall Officials: Marwa saad, MSc, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No